CLINICAL TRIAL: NCT01228318
Title: Bone Loss and Immune Reconstitution in HIV/AIDS (BLIR-HIV)
Acronym: BLIR-HIV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Ighovwerha Ofotokun, Associate Professor of Medicine, Emory University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00038739; BLIR-HIV (Other: Other)
Record Dates: First submitted 2010-10-23; First posted 2010-10-26 (Estimated); Results first posted 2018-06-26 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-05

CONDITIONS: HIV Infection; Bone Loss; Osteopenia; Osteoporosis
Keywords: HAART; Antiresorptive drugs; HIV/AIDS; Bone loss
MeSH Terms: conditions — HIV Infections; Bone Diseases, Metabolic; Osteoporosis; Acquired Immunodeficiency Syndrome | interventions — Zoledronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Zoledronic acid (Experimental): Subjects in this arm will receive 5 milligram (mg) per 100 milliliter (mL) solution of zoledronic acid infused intravenously over 15-30 minutes under the supervision of study personnel.
  Interventions: Drug: Zoledronic acid
- Placebo (Placebo Comparator): Subjects in the placebo arm will receive placebo containing 220 mg mannitol and 24 mg sodium citrate in a 100 mL ready-to-infuse solution administered iv over 15-30 minutes under the supervision of study personnel.
  Interventions: Drug: Zoledronic acid

INTERVENTIONS:
Drug: Zoledronic acid — 1. A single dose of reclast containing 5 mg/100 mL ready-to-infuse zoledronic acid solution administered over 15-30 minutes.
  2. A single dose of placebo containing 220 mg mannitol and 24 mg sodium citrate in a 100 mL ready-to-infuse solution, administered over 15-30 minutes.
  Other Names: Reclast

SUMMARY:
With the increasing age of people living with HIV/AIDS, age-induced osteoporosis is likely to be compounded by HIV/AIDS and HAART-associated bone loss. Mechanistically, osteoclasts the cells responsible for bone resorption form under the influence of the key osteoclastogenic cytokine receptor activator of nuclear factor kappa-Β ligand (RANKL). The osteoclastogenic and proresorptive activities of RANKL are moderated by its physiological decoy receptor osteoprotegerin (OPG). Imbalance in the ratio of RANKL to OPG alters osteoclastic bone resorption and lead to osteoporosis. Activated T- and B-cells are a major source of RANKL, while normal physiological B-cells are a major source of OPG. T-cells regulate the production of OPG by B-cells. Thus changes in the immune system induced by HIV/AIDS and/or by HAART could affect B-cell and T-cells RANKL and OPG production. Indeed, data from our group shows that in an animal model of HIV/AIDS, the HIV-1 Transgenic rat, the development of osteoporosis is recapitulated as observed in HIV-infected patients, and B-cell OPG and RANKL production are concurrently down regulated and upregulated respectively. Furthermore, preliminary data in HIV-infected subjects suggests dramatic acute upswing in bone resorption following HAART initiation that peaks at 12 weeks and then declines. Based on these findings, the investigators hypothesize HAART associated bone loss is driven by immune reconstitution. Because this effect of HAART is dramatic in magnitude but short in duration, the investigators propose to apply antiresorptive agent (zoledronic acid, reclast®) to specifically spare patients from this dramatic but acute bone damage.

DETAILED DESCRIPTION:
In a prospective, blinded placebo-controlled randomized trial, treatment naïve HIV-infected subjects initiating HAART will be assigned to HAART + zoledronic acid or HAART + placebo. Serial assessment of serum levels of bone markers, cellular expression of OPG/RANKL and other cytokines, cellular immune activation markers, serum bone regulating hormones, and bone mineral density (BMD) by dual-energy X-ray absorptiometry (DXA) scan will be undertaken at pre-defined time points from baseline through week 144 of HAART.

In the primary analysis, changes in serum C-Terminal Telopeptide (CTx) level, BMD, and cellular OPG/RANKL expression from baseline through week 24 will be quantitated and subsequently compared between treatment arms. In addition, the impact of zoledronic acid administration on these covariates will be assessed at various study time points. The relationship between OPG/RANKL expression, immune activation, serum bone regulating hormonal levels, and bone turnover will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 infection, as documented by any licensed serologic test and confirmed by a western blot or by a positive plasma HIV-1 RNA performed by any laboratory that has a Clinical Laboratory Improvement Amendments (CLIA) certification.
2. Meets Grady Infectious Disease Program (IDP) clinical criteria for antiretroviral therapy initiation, and subject and his/her provider are agreeable to subject initiating therapy with a regimen consisting of atazanavir (ATV)/ritonavir (RTV) + emtricitabine (FTC)/tenofovir (TDF) as part of his/her routine HIV management.
3. Ambulatory men and women age ≥ 30 ≤ 50 years.
4. Ability and willingness of subject or legal guardian/representative to give written informed consent.
5. Antiretroviral (ARV) drug-naïve (defined as ≤ 10 days of antiretroviral therapy (ART) at any time prior to entry).
6. Screening HIV-1 RNA ≥ 1000 copies/mL obtained within 90 days prior to study entry by any FDA-approved test for quantifying HIV-1 RNA at any laboratory that has a CLIA certification.
7. Laboratory values obtained within 90 days prior to study entry.

   * Absolute neutrophil count (ANC) ≥ 500/mm3
   * Hemoglobin ≥ 8.0 g/dL
   * Platelet count ≥ 40,000/mm3
   * Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase ≥ 3 x upper limit of normal (ULN)
   * Total bilirubin ≥ 2.5 x ULN
   * Calcium ≥ 8.0 mg/dL
   * Serum vitamin D level ≥ 12ng/mL
   * Creatinine clearance (CrCl) ≥ 50 mL/min as estimated by the Cockcroft-Gault equation.
8. Absence of history of non-HIV related active immunological or bone disorders such as:

   * Bone marrow or organ transplantation
   * Inflammatory bowel disease (ulcerative colitis, Crohn's disease)
   * Multiple Myeloma
   * Osteogenesis imperfecta
   * Osteomalacia
   * Osteosarcoma
   * Paget's disease
   * Postmenopausal osteoporosis
   * Rheumatoid arthritis
   * Systemic lupus erythematosus
   * Thyroid disorders (hyper/hypothyroidism)
9. Contraception requirements

   1. Female Subjects of Reproductive Potential:

      Female subjects of reproductive potential, who are participating in sexual activity that could lead to pregnancy, must agree to use at least one reliable method of contraception while participating in the study. Acceptable methods of contraception include:
      * Condoms (male or female) with or without a spermicidal agent
      * Diaphragm or cervical cap with spermicide
      * Intrauterine device (IUD)
      * Hormone-based contraceptive (must contain at ≥ 35 mcg of ethinyl estradiol)
   2. Female Subjects Who Are Not of Reproductive Potential.

Exclusion Criteria:

1. Pregnancy or breast feeding
2. Physical or biochemical evidence or a medical history of malignancy.
3. Currently (within the past 8 weeks) taking any medication with known influence on the immune or skeletal system (e.g. immune modulation therapy, glucocorticoids, steroid hormones, other bisphosphonates).
4. Osteoporosis defined as T-score <-2.5 at the hip, or spine, or history of osteoporotic fracture.
5. Prior or current use of zoledronic acid (reclast®)
6. Recent (within the past 6 months) or planned (within the next 6 months) invasive dental procedure.
7. Known allergy/sensitivity to study drugs or their formulations or mammalian cell derived drug products.
8. Any condition that, in the opinion of the investigators, would compromise the subject's ability to participate in the study.
9. Serious illness requiring systemic treatment and/or hospitalization until subject either completes therapy or is clinically stable on therapy, in the opinion of the investigators, for at least 7 days prior to study entry.
10. Requirement for any current medications that are prohibited with any study drugs. Prohibited medications must be discontinued at least 30 days prior to entry.
11. Current imprisonment or involuntary incarceration in a medical facility for psychiatric or physical illness.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2011-01; Primary Completion 2017-04-13 (Actual); Study Completion 2017-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Igho Ofotokun, MD, MSc, Principal Investigator — Emory University; Mervyn N Weitzmann, PhD, Principal Investigator — Emory University
Locations (1):
- Grady Infectious Diseases Clinic (Ponce Center), Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Vikulina T, Fan X, Yamaguchi M, Roser-Page S, Zayzafoon M, Guidot DM, Ofotokun I, Weitzmann MN. Alterations in the immuno-skeletal interface drive bone destruction in HIV-1 transgenic rats. Proc Natl Acad Sci U S A. 2010 Aug 3;107(31):13848-53. doi: 10.1073/pnas.1003020107. Epub 2010 Jul 19. PMID 20643942
- [Background] Ofotokun I, Weitzmann MN. HIV-1 infection and antiretroviral therapies: risk factors for osteoporosis and bone fracture. Curr Opin Endocrinol Diabetes Obes. 2010 Dec;17(6):523-9. doi: 10.1097/MED.0b013e32833f48d6. PMID 20844427
- [Result] Ofotokun I, Titanji K, Lahiri CD, Vunnava A, Foster A, Sanford SE, Sheth AN, Lennox JL, Knezevic A, Ward L, Easley KA, Powers P, Weitzmann MN. A Single-dose Zoledronic Acid Infusion Prevents Antiretroviral Therapy-induced Bone Loss in Treatment-naive HIV-infected Patients: A Phase IIb Trial. Clin Infect Dis. 2016 Sep 1;63(5):663-671. doi: 10.1093/cid/ciw331. Epub 2016 May 18. PMID 27193748
- [Derived] Ofotokun I, Collins LF, Titanji K, Foster A, Moran CA, Sheth AN, Lahiri CD, Lennox JL, Ward L, Easley KA, Weitzmann MN. Antiretroviral Therapy-Induced Bone Loss Is Durably Suppressed by a Single Dose of Zoledronic Acid in Treatment-Naive Persons with Human Immunodeficiency Virus Infection: A Phase IIB Trial. Clin Infect Dis. 2020 Oct 23;71(7):1655-1663. doi: 10.1093/cid/ciz1027. PMID 31621838

RESULTS

PARTICIPANT FLOW:
Recruitment Details: At the Grady Hospital Infectious Disease Clinic 343 subjects were assessed for eligibility and 280 were excluded. 63 viremic treatment-naïve adult HIV-infected subjects were randomized in a double-blinded, placebo-controlled study (ART+placebo N=29; ART+Zoledronic acid N=34). Participants were enrolled between January 2011 and August 2014.
Groups:
- Zoledronic Acid: Participants in this arm received a 5 milligrams (mg)/100 milliliter (mL) solution of zoledronic acid infused intravenously over 15-30 minutes under the supervision of study personnel.
  Study visits occurred at 12, 24, 48, 96, and 144 weeks.
- Placebo: Participants in the placebo arm received a placebo to match the study drug, containing 220 mg mannitol and 24 mg sodium citrate in a 100 mL ready-to-infuse solution administered intravenously over 15-30 minutes under the supervision of study personnel.
  Study visits occurred at 12, 24, 48, 96, and 144 weeks.
Period: Overall Study
Arm/Group | Zoledronic Acid | Placebo
Started | 34 | 29
Completed | 30 | 22
Not Completed | 4 | 7
Not completed — Clinic no show to receive intervention | 1 | 0
Not completed — Unable to contact | 2 | 5
Not completed — Moved | 0 | 2
Not completed — Incarcerated | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Zoledronic Acid: Participants in this arm received a 5mg/100mL solution of zoledronic acid infused intravenously over 15-30 minutes under the supervision of study personnel.
- Placebo: Participants in the placebo arm received a placebo to match the study drug, containing 220 mg mannitol and 24 mg sodium citrate in a 100 mL ready-to-infuse solution administered intravenously over 15-30 minutes under the supervision of study personnel.
- Total: Total of all reporting groups
Arm/Group | Zoledronic Acid | Placebo | Total
Number analyzed (Participants) | 34 | 29 | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 34 | 29 | 63
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 23 | 50
  Male | 7 | 6 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 32 | 29 | 61
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 27 | 26 | 53
  White | 7 | 3 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 34 | 29 | 63
Body Mass Index (BMI) [Median (Full Range); unit: kg/m^2] | 24.4 [18.9 to 41.2] | 23.8 [16.9 to 38.7] | 23.8 [16.9 to 41.2]
Cluster of differentiation 4 (CD4) T-cell count [Median (Full Range); unit: cells/uL] | 91.5 [5 to 239] | 117 [3 to 574] | 101 [3 to 574]
HIV-1 Viral Load [Median (Full Range); unit: log10 copies/ml] | 4.97 [3.69 to 6.44] | 4.93 [2.51 to 6.06] | 4.96 [2.51 to 6.44]
Weight [Median (Full Range); unit: kilograms] | 72.9 [49.8 to 118.2] | 73.3 [54.9 to 107.2] | 73.3 [49.8 to 118.2]
Age [Median (Full Range); unit: years] | 38 [30 to 50] | 37 [30 to 51] | 38 [30 to 51]
Height [Median (Full Range); unit: inches] | 69 [61 to 76] | 70 [61 to 77] | 70 [61 to 77]

OUTCOME MEASURES:

1. Primary Outcome: Baseline-Adjusted Means for C-terminal Telopeptide of Collagen (CTx) Levels
Description: Serum C-terminal telopeptide of collagen (CTx) levels through week 144 were examined by evaluating the baseline-adjusted means. The baseline-adjusted CTx mean is defined as the predicted response value obtained by fitting the regression equation for each treatment arm at the mean baseline value for the 2 treatment arms. The adjusted means were estimated using analysis of covariance at each scheduled clinical visit. The expected outcome is that HIV-infected individuals will display increased indices of bone resorption (CTx) as a result of diminished bone mineral density (BMD). Lower CTx values indicate that better maintenance of bone mineral density.
Time Frame: Baseline, Week 12 through Week 144
Population: Participants with CTx measurements at the indicated week are included in this analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: ng/ml
Groups:
- Zoledronic Acid: Subjects in this arm will receive 5mg/100mL solution of zoledronic acid infused intravenously over 15-30 minutes under the supervision of study personnel.
  Zoledronic acid: a. A single dose of reclast containing 5 mg/100 mL ready-to-infuse zoledronic acid solution administered over 15-30 minutes.
  b. A single dose of placebo containing 220 mg mannitol and 24 mg sodium citrate in a 100 mL ready-to-infuse solution, administered over 15-30 minutes.
- Placebo: Subjects in the placebo arm will receive placebo containing 220 mg mannitol and 24 mg sodium citrate in a 100 mL ready-to-infuse solution administered iv over 15-30 minutes under the supervision of study personnel.
  Zoledronic acid: a. A single dose of reclast containing 5 mg/100 mL ready-to-infuse zoledronic acid solution administered over 15-30 minutes.
  b. A single dose of placebo containing 220 mg mannitol and 24 mg sodium citrate in a 100 mL ready-to-infuse solution, administered over 15-30 minutes.
Arm/Group | Zoledronic Acid | Placebo
Number analyzed (Participants) | 31 | 26
ng/ml
  Week 12: number analyzed (Participants) | 30 | 26
  Week 12 | 0.092 [0.040 to 0.145] | 0.297 [0.240 to 0.353]
  Week 24: number analyzed (Participants) | 31 | 25
  Week 24 | 0.122 [0.074 to 0.171] | 0.331 [0.276 to 0.384]
  Week 48: number analyzed (Participants) | 28 | 24
  Week 48 | 0.122 [0.077 to 0.168] | 0.264 [0.215 to 0.313]
  Week 72: number analyzed (Participants) | 25 | 22
  Week 72 | 0.138 [0.088 to 0.189] | 0.242 [0.188 to 0.296]
  Week 96: number analyzed (Participants) | 23 | 23
  Week 96 | 0.126 [0.042 to 0.209] | 0.321 [0.238 to 0.404]
  Week 120: number analyzed (Participants) | 20 | 20
  Week 120 | 0.137 [0.088 to 0.187] | 0.201 [0.151 to 0.250]
  Week 144: number analyzed (Participants) | 21 | 20
  Week 144 | 0.148 [0.096 to 0.200] | 0.200 [0.147 to 0.254]

2. Secondary Outcome: Baseline-Adjusted Means of Osteocalcin
Description: Osteocalcin was evaluated to examine the inhibitory effect of single dose zoledronic acid on HAART associated changes in markers of bone turnover. Osteocalcin is released from bone during resorption and higher levels in the circulatory system indicate increased bone turnover. HIV-infected individuals are expected to have increased bone resorption. The baseline-adjusted osteocalcin mean is defined as the predicted response value obtained by fitting the regression equation for each treatment arm at the mean baseline value for the 2 treatment arms. The adjusted means were estimated using analysis of covariance at the Week 144 clinic visit. Baseline-adjusted means of osteocalcin at week 144 are presented.
Time Frame: Baseline, Week 144
Population: Participants with osteocalcin measurements at Week 144 are included in this analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: ng/ml
Arm/Group | Zoledronic Acid | Placebo
Number analyzed (Participants) | 21 | 20
ng/ml | 9.176 [4.557 to 13.796] | 13.597 [8.862 to 18.332]

3. Other Pre Specified Outcome: Baseline-Adjusted Means of Dual-energy X-ray Absorptiometry (DXA)
Description: Development of osteoporosis was assessed by examining bone mineral density (BMD) by DXA scan. Baseline-adjusted means of DXA scan Z-scores are presented for the lumbar spine (L1-L4), left hip, and femur neck. The baseline-adjusted BMD mean is defined as the predicted response value obtained by fitting the regression equation for each treatment arm at the mean baseline value for the 2 treatment arms. The adjusted means were estimated using analysis of covariance at the Week 144 clinic visit. Bone density Z-scores tell how close to the average that a person is (adjusted for age, race, and gender). A Z-score of 0 means the value matches that of the average person. Z-score values below 0 indicate lower than average bone density while values above 0 indicate higher bone density than the average person.
Time Frame: Baseline, Week 144
Population: This analysis includes participants who had a DXA scan performed at baseline and at least one additional study visit.
Measure: Least Squares Mean (95% Confidence Interval); unit: Z score
Arm/Group | Zoledronic Acid | Placebo
Number analyzed (Participants) | 29 | 20
Z score
  Lumbar Spine | -0.177 [-0.371 to 0.016] | -0.836 [-1.062 to -0.609]
  Hip | -0.860 [-0.992 to -0.728] | -1.092 [-1.246 to -0.938]
  Femoral Neck | -0.665 [-0.833 to -0.498] | -0.817 [-1.012 to -0.622]

4. Post Hoc Outcome: Percentage of Participants With Virological Suppression by Week 144
Description: The percentage of participants achieving viral load suppression by study week 144. Virologic suppression was defined as HIV RNA polymerase chain reaction (PCR) (viral loads) less than 50 copies per mL.
Time Frame: Week 144
Population: All participants are included in this analysis, using all available measurements of viral load.
Measure: Number; unit: percentage of participants
Arm/Group | Zoledronic Acid | Placebo
Number analyzed (Participants) | 34 | 29
percentage of participants | 91 | 100

5. Post Hoc Outcome: CD4 T Cell Count
Description: Immunologic response measured by CD4 T cell count by treatment arm and weeks on study.
Time Frame: Baseline, Week 144
Population: This analysis includes participants with a CD4 count measurement at the time points indicated.
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Zoledronic Acid | Placebo
Number analyzed (Participants) | 34 | 29
cells/uL
  Baseline | 102 (69) | 155 (145)
  Week 144: number analyzed (Participants) | 31 | 22
  Week 144 | 347 (27) | 439 (52)

ADVERSE EVENTS:
Time Frame: Adverse effects elicited from the BLIR patient at each scheduled visit (12, 24, 48, 96, and 144 weeks) using the Case Report Form Checklist of 36 HAART Signs and Symptoms. Participants were also volunteered complaints of side effects that were outside of the checklist.
Description: The definition of adverse event and/or serious adverse event, used to collect adverse event information, does not differ from the ClinicalTrials.gov definitions.
Arm/Group | Zoledronic Acid | Placebo
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/29
Serious Adverse Events (participants affected / at risk) | 7/34 | 6/29
Other Adverse Events (participants affected / at risk) | 34/34 | 28/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zoledronic Acid (N=34) | Placebo (N=29)
Hospitalization due to pancreatitis (Endocrine disorders) | 1 (1) | 0 (0)
Hospitalization due to abdominal pain (General disorders) | 1 (1) | 0 (0) — Participant was hospitalized with complaints of abdominal pain and was discharged after being observed for 24 hours.
Hospitalization due to community acquired pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Hospitalization due to neurosyphilis (Infections and infestations) | 1 (1) | 0 (0)
Hospitalization (General disorders) | 1 (1) | 0 (0) — Participant was admitted with multiple diagnoses that were unrelated to study treatment
Hospitalization due to gastro esphageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) — Participant was admitted due to chest pain and abnormal electrocardiogram; cardiac tests were normal and gastro esophageal reflux disease was diagnosed
Psychiatric hospitalization (Psychiatric disorders) | 0 (0) | 1 (1) — Participant admitted to psychiatric unit due to homicidal intentions against family member. This event is considered unrelated to study treatment.
Hospitalization due to brochitis and otitis externa (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hospitalization related to Graves' Disease (Endocrine disorders) | 0 (0) | 1 (3)
Hospitalization due to sub-acute cerebrovascular accident (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zoledronic Acid (N=34) | Placebo (N=29)
Fatigue (General disorders) | 28 (176) | 22 (145)
Cough (Respiratory, thoracic and mediastinal disorders) | 28 (141) | 22 (79)
Nasal/sinus drainage (Respiratory, thoracic and mediastinal disorders) | 28 (141) | 22 (79)
Diarrhea (Gastrointestinal disorders) | 26 (113) | 18 (69)
Night sweats (General disorders) | 26 (87) | 15 (56)
Headache (General disorders) | 26 (110) | 15 (81)
Numbness/tingling (General disorders) | 27 (156) | 13 (114)
Rash (head, shoulder, feet) (Skin and subcutaneous tissue disorders) | 21 (90) | 18 (76)
Decreased libido (General disorders) | 24 (127) | 15 (92)
Flatulence (Gastrointestinal disorders) | 24 (128) | 13 (91)
Depression (Psychiatric disorders) | 21 (150) | 16 (131)
Weight loss (General disorders) | 21 (46) | 15 (42)
Loss of appetite (General disorders) | 20 (66) | 15 (63)
Insomnia (General disorders) | 21 (140) | 14 (90)
Myalgias (General disorders) | 20 (99) | 15 (89)
Arthralgias (General disorders) | 18 (71) | 17 (105)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 20 (101) | 13 (94)
Flulike symptoms (General disorders) | 18 (31) | 13 (19)
Fever (General disorders) | 15 (26) | 15 (22)
Chills (General disorders) | 17 (29) | 13 (27)
Nausea (General disorders) | 17 (55) | 13 (45)
Dyspepsia (Gastrointestinal disorders) | 16 (42) | 13 (34)
Blurred vision (General disorders) | 17 (76) | 12 (93)
Loss of memory (General disorders) | 15 (99) | 12 (83)
Abdominal pain (General disorders) | 13 (36) | 9 (45)
Vomiting (Gastrointestinal disorders) | 10 (20) | 10 (20)
Motor weakness (General disorders) | 11 (32) | 9 (78)
Asthenia (General disorders) | 10 (33) | 9 (62)
Dysphagia (Gastrointestinal disorders) | 7 (29) | 8 (25)
Oral thrush (Infections and infestations) | 9 (11) | 6 (14)
Oral pain (General disorders) | 8 (16) | 6 (20)
Photophobia (General disorders) | 4 (18) | 10 (37)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 6 (9)
Bone pain (General disorders) | 6 (28) | 5 (30)
Vein distended (Vascular disorders) | 2 (15) | 3 (17)
Odynophagia (General disorders) | 1 (1) | 1 (1)
Kaposi sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (10) | 0 (0)
Dizziness (General disorders) | 5 (10) | 4 (12)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (6)
Chest pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (8)
Back pain (General disorders) | 7 (36) | 5 (19)
Tooth ache (General disorders) | 3 (46) | 4 (42)
Tinnitus (Ear and labyrinth disorders) | 2 (15) | 2 (9)
Generalized muscle pain (General disorders) | 2 (3) | 2 (9)
Left eye twitching (General disorders) | 2 (2) | 1 (3)
Pain from shingles (Infections and infestations) | 2 (6) | 1 (3)
Anxiety (Psychiatric disorders) | 1 (6) | 1 (4)
Bloody stool (Gastrointestinal disorders) | 2 (3) | 0 (0)
Dry mouth (General disorders) | 0 (0) | 2 (7)
Groin pain (Reproductive system and breast disorders) | 2 (3) | 0 (0)
Muscle cramps (hands, feet, legs) (Musculoskeletal and connective tissue disorders) | 5 (8) | 1 (1)
Intermittent nose bleed (General disorders) | 2 (3) | 0 (0)
Pain in right ear (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Foot pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 3 (5)
Throat pain (General disorders) | 0 (0) | 2 (2)
Abdominal tenderness (General disorders) | 0 (0) | 1 (2)
Anal pain (General disorders) | 1 (1) | 0 (0)
Ankle tenderness/pain (Musculoskeletal and connective tissue disorders) | 1 (3) | 1 (1)
Arm pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Flank pain (General disorders) | 3 (8) | 0 (0)
Bitter mouth taste (Gastrointestinal disorders) | 2 (9) | 0 (0)
Bladder spasms (Renal and urinary disorders) | 0 (0) | 1 (2)
Bloating (General disorders) | 0 (0) | 1 (1)
Boil left buttock (Infections and infestations) | 0 (0) | 1 (1)
Bone pain in left hand (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bruising easily (General disorders) | 0 (0) | 1 (1)
Bump inside mouth (General disorders) | 0 (0) | 1 (1)
Burning in chest with excertion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Constipation (Gastrointestinal disorders) | 1 (2) | 0 (0)
Dark spots (Skin and subcutaneous tissue disorders) | 3 (10) | 0 (0)
Dark urine (Renal and urinary disorders) | 1 (4) | 0 (0)
Decreased hearing/ear stopped up (Ear and labyrinth disorders) | 2 (4) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (5) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Easily distracted (General disorders) | 1 (7) | 0 (0)
Entire body heat (General disorders) | 1 (1) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Itchy/watery eye (Eye disorders) | 1 (1) | 3 (7)
Facial acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Frequent urination (Renal and urinary disorders) | 1 (3) | 0 (0)
General body aches (General disorders) | 0 (0) | 1 (1)
Hair thinning (General disorders) | 0 (0) | 1 (2)
Hearing voices (Psychiatric disorders) | 0 (0) | 1 (5)
Herpes outbreak (Infections and infestations) | 0 (0) | 2 (4)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0)
Hotflashes (General disorders) | 2 (12) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Knee swollen (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lower extremity edema (Blood and lymphatic system disorders) | 2 (4) | 1 (1)
Lower left leg pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Left sided weakness (General disorders) | 0 (0) | 1 (2)
Numbness (hands, legs, body) (General disorders) | 3 (4) | 1 (1)
Loss of balance (General disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain/stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (11)
Pain in right knee (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rash left forehead (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Right shoulder discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Right facial swelling (General disorders) | 0 (0) | 1 (1)
Right side weakness (General disorders) | 0 (0) | 1 (9)
Right wrist pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Salivation (General disorders) | 1 (8) | 0 (0)
Scalp pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Seeing spots (Eye disorders) | 0 (0) | 2 (4)
Stomach feels tight (General disorders) | 1 (3) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 1 (3)
Urinary retention (Renal and urinary disorders) | 1 (4) | 0 (0)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 1 (1)
Vaginal itching (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Welts when skin scratched (Skin and subcutaneous tissue disorders) | 2 (10) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This single site proof-of-concept phase 2b study had a small sample size & a 144-week study duration so it could not evaluate the impact of the intervention on long-term bone outcomes. The population enrolled limited the generalization of findings.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2014-06-06): https://cdn.clinicaltrials.gov/large-docs/18/NCT01228318/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2014-06-25): https://cdn.clinicaltrials.gov/large-docs/18/NCT01228318/Prot_SAP_001.pdf